CLINICAL TRIAL: NCT01158612
Title: The Effect of Local Injectet GH on the Collagen Synthesis in the Ligamentum Patella
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2-2010-039
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Growth Hormone; Elderly
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Growth hormone (Experimental): The effect of Growth hormone on the collagen synthesis rate
  Interventions: Drug: Growth Hormone
- Saline (Placebo Comparator)
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone — infusion of Growth hormone in the patella tendon.
  Other Names: infusion of Saline in the patella tendon.

SUMMARY:
Tendon and ligament injuries are a frequent problem among athletes but also in the general population. The healing process is a prolonged process, and complete recovery of tissue strength is nearly never reached. The purpose of this study is to examine the effect of local injection of human Growth Hormone on tendon collagen synthesis.

DETAILED DESCRIPTION:
Tendon and ligament injuries are a frequent problem among athletes but also in the general population. The healing process is a prolonged process, and complete recovery of tissue strength is nearly never reached. The purpose of this study is to examine the effect of local injection of human Growth Hormone on tendon collagen synthesis.

in order to investigate the collagen synthesis potential and the influence of growth hormone, 12 elderly males age > 50 year, is enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25.0

Exclusion Criteria:

* earlier knee injury

Ages: 55 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
• Fraktionele collagen protein synthesis in human patella tendon | 01122010

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, PH.D., Principal Investigator
Locations (1):
- Århus universitetshospital nørrebrogade 44, Århus C, Denmark